CLINICAL TRIAL: NCT02585219
Title: Pilot Feasibility of 11C-MET-PET as a Post-surgery Baseline Scan in the Follow-up of High-grade Gliomas for the Detection of Tumor Recurrence.
Brief Title: Pilot Viability of 11C-MET-PET as a Post-surgery Baseline Scan in High-grade Gliomas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Ronald W J van Rheenen, MD, Nuclear Medicine Physician, University Medical Center Groningen
Other Study IDs: NL50485.042.14
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High-grade Glioma Patients: Patients with suspicion of newly diagnosed high-grade glioma eligible for standard therapy (surgical resection followed by chemoradiotherapy).
  Patients with a second brain tumor, brain surgery earlier or prior radiotherapy to the brain are excluded. Patients with only a biopsy be excluded.
  The group will consist of 10 patients. This number may be adjusted for patients who are found to have a different diagnosis after histological examination or fall out. For a pilot feasibility study our experience that a number of 10 patients is sufficient for PET examination.

SUMMARY:
The tracer 11C-methionine (11 C-MET) is used as a specific cell proliferation tracer which shows metabolically active tumordeposities. A healthy brain barely takes up 11C-MET, causing the difference between the background and the tumor to be realively high. In addition, there is relatively little 11C-MET uptake in inflammatory processes. This makes 11C-MET a very suitable positron emission tomography (PET) tracer in order to differentiate between tumor progression and therapy changes. The latter is a major clinical problem for which further investigation is necessary.

In order to be able to make this differentiation, a direct post-operative baseline scan is required. With regard to the advanced MRI sequences, it is known that it is necessary to produce the post-operative baseline scan within 48 hours. After that timeframe, operation induced changes start to occur, such as granulation tissue. In that case the interpretation of the scan is no longer possible. Immediately postoperatively (<48 hours) 11C-MET has never been used before. Therefore, it is unknown whether 11C-MET provides a good baseline scan directly after surgery. This pilot will investigate the feasibility of this 11C-MET baseline scan and comparison the results with the advanced MRI sequences.

DETAILED DESCRIPTION:
Conventional MRI, advanced MRI and 11C-MET-PET will be conducted on the same day. The advanced MRI will consist of diffusion weighted imaging (DWI), perfusion imaging by contrast technique (DSC) and spectroscopy (MRS). The post-operative MRI and PET scan will be produced within 48 hours after surgery (with the aim that operative effects are not visible on the baseline scan). This corresponds to the current practice of conventional MRI follow-up at the end of the radiotherapy.

The comparison with the pre-operative scan is to assess the viability of the post-operative scan. It will assessed whether the preoperative tumor uptake will disappear in accordance to the resection, as shown by the advanced MRI sequences. In addition, it will be assessed whether there are no interfering postoperative effects. The 11C-MET-PET scans will be interpreted in comparison with the quantitative results obtained with advanced MRI sequences (perfusion / diffusion / oxygenation / spectroscopy). If an immediate postoperative 11C-MET-PET proves to be feasible, than this will provide a basis for further research. This future research consist out of the differentiation between tumor progression and therapy change, one of the most urgent clinical dilemmas in neuro-oncology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of newly diagnosed high-grade glioma who qualify for the standard treatment. Written informed consent

Exclusion Criteria:

* Patients with recurrent high-grade glioma or other brain tumor as a secondary diagnosis are excluded.
* In addition, all patients who have had previous brain surgery or radiotherapy to the brain are also excluded.
* Patients with only a biopsy will be excluded. Patients under the age of 18 years will not be included.
* General exclusion criteria for MRI are exclusion criteria for participation in this study. The general MRI exclusion criteria are: not MRI compatible ferromagnetic material, pregnancy (or presumption thereof) and claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of newly diagnosed high-grade glioma eligible for standard therapy (surgical resection followed by chemoradiotherapy).
  Patients with a second brain tumor, brain surgery earlier or prior radiotherapy to the brain are excluded. Patients with only a biopsy be excluded.
  The group will consist of 10 patients. This number may be adjusted for patients who are found to have a different diagnosis after histological examination or fall out. For a pilot feasibility study our experience that a number of 10 patients is sufficient for PET examination.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Visual comparison of pre- and post-surgery 11C-MET-PET | 1 week between pre- and post-surgery 11C-MET-PET
  The 11C-MET-PET within 48 hours postoperatively will be assessed visually and quantitatively and compared with the preoperative 11C-MET-PET scan. The 11C-MET-PET data will also be checked by comparison with the results of the advanced MRI sequences. Specifically the comparison will include evaluation of surgical success (all former positive 11C-MET uptake removed) and evaluation of possible post-surgical effects on the second 11C-MET-PET.